CLINICAL TRIAL: NCT04727996
Title: Phase II Study of Sitravatinib in Combination With Tislelizumab in Patients With Advanced Biliary Tract Cancer Who Have Failed to At Least 1 Prior Systemic Treatment
Brief Title: Phase II Study of Sitravatinib in Combination With Tislelizumab in Patients With Advanced Biliary Tract Cancer
Acronym: BTC-BGB
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Principal Investigator, Do-Youn Oh, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2005-156-1126
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Advanced Biliary Tract Cancer
MeSH Terms: interventions — sitravatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sitravatinib/Tislelizumab (Experimental): All patients will receive sitravatinib 120 mg orally once daily in combination with tislelizumab 200 mg IV once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Sitravatinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Sitravatinib — 120 mg will be administered orally once daily
  Other Names: MGCD516
Drug: Tislelizumab — 200 mg will be administered intravenously (IV) once every 3 weeks
  Other Names: BGB-A317

SUMMARY:
This is open-label, phase II study enrolling advanced BTC patients who have failed to 1st-line chemotherapy.

DETAILED DESCRIPTION:
<Study Objectives>

Primary Objectives:

To characterize the efficacy of Sitravatinib and Tislelizumab combination in biliary tract cancer patients who have failed to 1st-line chemotherapy but no more than 2 lines of prior chemotherapy regimen

Secondary Objectives:

To see the safety of Sitravatinib and Tislelizumab combination in biliary tract cancer patients who have failed to 1st-line chemotherapy

<Rationale> sitravatinib and tislelizumab may elicit greater antitumor activity, as sitravatinib is predicted to enhance several steps in the cancer immunity Cycle that may augment the efficacy of tislelizumab. First, the antitumor activity of sitravatinib may promote the release of tumor antigens. Second, inhibition of the split kinase receptors VEGFR-2 and KIT may decrease the number of Tregs and MDSCs, thus promoting the expansion and migration of antitumor cytotoxic T cells, and their infiltration into tumor tissue. Third, sitravatinib may reverse the immunosuppressive effects within the tumor microenvironment that are mediated by the TAM receptors through inhibition of MERTK, resulting in an increased number of M1- versus M2-polarized macrophages and release of IL 12, IL-6, and TNF. These downstream effects enhance CD8+ T-cell activation, and through the inhibition of AXL, promote increased antigen presentation through termination of the Toll-like receptor dependent inflammatory response in dendritic cells.

In biliary tract cancer, this sitravatinib and tislelizumab combination has not been tested so far. In this protocol, we will test sitravatinib and tislelizumab combination in advanced biliary tract cancer.

<hypothesis> Selective receptor tyrosine kinases inhibit key molecular and cellular pathways strongly implicated in checkpoint inhibitor resistance and therefore represent reasonable strategies to enhance or restore antitumor immunity when combined with anti-PD-1 or anti-PD-L1 monoclonal antibodies.

<Study design> This is open-label, phase II study enrolling advanced BTC patients who have failed to 1st-line chemotherapy.

All patients will receive sitravatinib 120 mg orally once daily in combination with tislelizumab 200 mg IV once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent and any locally-required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations 2. Age≥ 20 years at time of study entry 3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 4. Life expectancy of ≥ 16weeks 5. Histologically proven BTC, including intrahepatic cholangiocarcinoma, extrahepatic bile duct cancer, gallbladder cancer, ampulla of vater cancer 6. Unresectable or recurrent 7. Failed to 1st-line chemotherapy for their advanced BTC, but no more than 2 lines of prior chemotherapy regimen 8. At least one measurable lesion that can be accurately assessed at baseline by computed tomography (CT) (magnetic resonance imaging [MRI] where CT is contraindicated) and is suitable for repeated assessment as per RECIST 1.1.

  9. Body weight >30kg 10. Adequate normal organ and marrow function measured within 28 days prior to administration of study treatment as defined below:

  • Haemoglobin ≥9.0 g/dL

  • Absolute neutrophil count (ANC) ≥ 1.5 x 10 9/L
  * Platelet count ≥ 75 x 10 9/L
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN), or estimated glomerular filtration rate ≥ 60 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equation
  * AST and ALT ≤ 3.0 x ULN, or AST and ALT ≤ 5.0 x ULN for patients with documented liver metastases
  * Serum total bilirubin ≤ 1.5 x ULN (total bilirubin must be < 3 x ULN for patients with Gilberts syndrome)
  * International normalized ratio (INR) ≤ 1.5 or prothrombin time ≤ 1.5 x ULN
  * Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN

    11. Patients with inactive/asymptomatic carrier, chronic, or active hepatitis B virus (HBV) must have HBV deoxyribonucleic acid (DNA) < 500 IU/mL (or 2500 copies/mL) at Screening 12. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥ 120 days after the last dose of study drugs and have a negative serum pregnancy test ≤ 7 days of first dose of study drugs 13. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of study drugs

Exclusion Criteria:

* 1. Unacceptable toxicity on prior anti-PD-1/PD-L1 treatment, defined as follows:

  1. ≥ Grade 3 AE related to anti-PD-1/PD-L1 treatment that did not respond to standard therapy and warranted treatment discontinuation.
  2. ≥ Grade 2 irAE(immune-related adverse event) associated with anti-PD-1/PD-L1 unless the AE(adverse event) resolved or was well controlled by withholding the anti-PD-1/PD-L1 and/or treatment with steroids, with the exception of prior colitis, encephalitis, myocarditis, hepatitis, uveitis and pneumonitis, which are exclusionary.
  3. Central nervous system or ocular AE of any grade related to anti-PD-1/PD-L1 Note: Patients with a prior endocrine AE are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.

     2. Active leptomeningeal disease or uncontrolled, untreated brain metastasis

     • Patients with a history of treated and, at the time of screening, asymptomatic CNS metastases are eligible, provided they meet all the following:

  <!-- -->

  1. Brain imaging at screening shows no evidence of interim progression
  2. All brain metastases with supratentorial location
  3. No ongoing requirement for corticosteroids as therapy for CNS disease; anticonvulsants at a stable dose allowed
  4. No stereotactic radiation or whole-brain radiation within 14 days prior to first dose of study drug(s)

     * Patients with new asymptomatic central nervous system metastases detected at the screening scan must receive radiation therapy and/or surgery for central nervous system metastases.
  5. Following treatment, these patients may then be eligible, provided all other criteria, including those for patients with a history of brain metastases, are met.

     3. Active autoimmune diseases or history of autoimmune diseases that may relapse

     Note: Patients with the following diseases are not excluded and may proceed to further screening:
  6. Controlled Type I diabetes
  7. Hypothyroidism (provided it is managed with hormone replacement therapy only)
  8. Controlled celiac disease
  9. Skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, alopecia)
  10. Any other disease that is not expected to recur in the absence of external triggering factors 4. Any active malignancy ≤ 2 years before first dose of study drugs except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast) 5. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before first dose of study drugs

      Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:

  <!-- -->

  1. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent)
  2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
  3. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a non-autoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen) 6. Uncontrolled diabetes or > Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management or ≥ Grade 3 hypoalbuminemia ≤ 14 days before first dose of study drugs 7. History of interstitial lung disease, noninfectious pneumonitis or uncontrolled diseases, including pulmonary fibrosis, acute lung diseases, etc.

     8. Severe chronic or active infections (including tuberculosis infection, etc.) requiring systemic antibacterial, antifungal or antiviral therapy, within 14 days prior to first dose of study drugs 9. Known history of HIV infection 10. Active hepatitis C infection (defined by a detectable HCV RNA). 11. Any major surgical procedure requiring general anesthesia ≤ 28 days before first dose of study drugs 12. Prior allogeneic stem cell transplantation or organ transplantation 13. Any of the following cardiovascular risk criteria:

  <!-- -->

  1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days before first dose of study drugs
  2. Symptomatic pulmonary embolism ≤ 28 days before first dose of study drugs
  3. Any history of acute myocardial infarction ≤ 6 months before first dose of study drugs
  4. Any history of heart failure meeting New York Heart Association Classification III or IV ≤ 6 months before first dose of study drugs
  5. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before first dose of study drugs
  6. Any history of cerebrovascular accident ≤ 6 months before first dose of study drugs
  7. QTc interval (corrected by Fridericia's method) > 450 msec Note: If QTc interval is > 450 msec on initial electrocardiogram (ECG), a follow up ECG will be performed to confirm result
  8. Cardiac left ventricular ejection fraction ≤ 40% or lower limit of normal as assessed by echocardiography. The same modality used at baseline must be applied for subsequent evaluations.
  9. Any episode of syncope or seizure ≤ 28 days before first dose of study drugs 14. Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) 15. Hypersensitivity to tislelizumab or sitravatinib, to any ingredient in the formulation, or to any component of the container 16. Bleeding or thrombotic disorders or use of anticoagulants such as warfarin or similar agents requiring therapeutic INR monitoring within 6 months before first dose of study drugs 17. Any systemic chemotherapy within 28 days of the first dose of study drugs or immunotherapy (eg, interleukin, interferon, thymoxin, etc.), hormone therapy, targeted therapy, or any investigational therapies within 14 days or 5 half-lives (whichever is shorter) of first dose of study drugs 18. Any herbal medicine used to control cancer within 14 days of first dose of study drugs 19. Toxicities (as a result of prior anticancer therapy) that have not improved to baseline or stabilized, except for AEs not considered a likely safety risk (eg, alopecia, neuropathy, and specific laboratory abnormalities) 20. Administration of live vaccine ≤ 4 weeks prior to first dose of study drugs Note: Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.

     21. Underlying medical conditions or alcohol or drug abuse or dependence that will be unfavorable for the administration of study drugs or affect the explanation of drug toxicity or AEs; or expected insufficient compliance during the study according to investigator's judgement 22. Participation in another clinical study, unless it is an observational (non interventional) clinical study or during the follow-up period of an interventional study 23. Inability to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction 24. Spinal cord compression in one or more of the following criteria

  <!-- -->

  1. Not definitively treated with surgery and/or radiation
  2. Treated but without evidence that disease has been clinically stable for > 2 weeks prior to first dose of study drugs 25. Pregnant or breastfeeding woman 26. Regardless of the severity, patients with any signs or medical history of bleeding; within 4 weeks prior to allocation, patients with any bleeding events ≥ CTCAE level 3, unhealed wounds, ulcers or fractures 27. Patients with artery/venous thrombotic occurred within 6 months before allocation, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | every 6weeks
  To assess the efficacy of Sitravatinib and Tislelizumab combination on DCR (disease control rate) in biliary tract cancer patients who have failed to 1st-line chemotherapy

SECONDARY OUTCOMES:
overall response rate | every 6weeks
  Partial response and complete response
progression-free survival | every 6weeks
  Progression-free survival was defined as the duration between beginning of treatment and disease progression, any cause of death before disease progression, or the last follow-up.The event was defined as disease progression and any cause of death.
overall survival | every 3months
  Overall survival was measured from the randomization to the last follow-up or any cause of death. The event was defined as any cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, M.D., PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon J, Lee CK, Kim JW, Kang B, Park SJ, Kim JW, Chon HJ, Choi HJ, Lee MA, Kim TY, Oh DY. Open-label, single-arm, phase II trial to investigate the efficacy of sitravatinib plus tislelizumab combination as a second-line treatment for advanced biliary tract cancer. J Hepatol. 2025 Nov 24:S0168-8278(25)02626-1. doi: 10.1016/j.jhep.2025.10.032. Online ahead of print. PMID 41297674